CLINICAL TRIAL: NCT04914143
Title: A Prospective, Single Center, Randomized, Double-blind Clinical Study to Evaluate the Effect of Broken Ganoderma Lucidum Spore Powder on Quality of Life and Immune Function in Patients With Diffuse Large B-cell Lymphoma After Chemotherapy
Brief Title: the Effect of Broken Ganoderma Lucidum Spore Powder on Quality of Life and Immune Function in Patients With Diffuse Large B-cell Lymphoma After Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-261
Record Dates: First submitted 2021-06-01; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: broken Ganoderma lucidum spore powder
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: broken Ganoderma lucidum spore powder
- placebo comparator group (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: broken Ganoderma lucidum spore powder — The experimental group was treated with broken Ganoderma lucidum spore powder after chemotherapy
  Arms: Experimental group
Other: placebo — the control group was treated with placebo after chemotherapy
  Arms: placebo comparator group

SUMMARY:
The purpose of this study was to explore the effect of broken Ganoderma lucidum spore powder on improving the quality of life and immune recovery of patients after chemotherapy. Objective To observe the adjuvant treatment with broken wall Ganoderma lucidum spore powder in patients with diffuse large B-cell lymphoma after standard chemotherapy according to NCCN guidelines. To evaluate and compare the immunoglobulin (IGA, IgM, IgG), T cell subsets (CD3 +, CD4 +, CD8 +, CD4 + / CD8 +), Th1 / Th2 cytokine determination, quality of life score, leukocyte recovery rate, infection rate, infection rate To evaluate the effect of Ganoderma lucidum spore powder in improving the quality of life and immune function of patients after chemotherapy. At the same time, the liver and kidney function and adverse drug events were closely monitored during the study to explore the clinical safety of wall broken Ganoderma lucidum spore powder as adjuvant drug.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse large B-cell lymphoma，NOS
* all patients were diagnosed for the first time
* between 18-75 years old, male and female
* ECoG 0-3 ，the expected survival was more than 6 months
* the pregnancy test of women of childbearing age was negative; Male and female patients should agree to take effective contraceptive measures during the treatment period and one year of follow-up;
* sign the informed consent before the test screening

Exclusion Criteria:

* those who are known to be allergic to the study drug or its related components; Or allergic patients
* uncontrolled psychosis
* participating in other trials at the same time, and using experimental drugs that may affect the efficacy and safety evaluation
* impairment of liver and kidney function
* HIV antibody positive;
* HBsAg positive hepatitis B carriers and confirmed hepatitis B and C patients;
* pregnant or lactating women and patients who do not agree to take effective contraceptive measures;
* the patient is unable to swallow the capsule or has a disease or condition that seriously affects the gastrointestinal function;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Detection of immunoglobulin (IGA, IgM, IgG) | half a year
T cell subsets | half a year
  T cell subsets (CD3 +, CD4 +, CD8 +, CD4 + / CD8 +)
Th1 / Th2 cytokines | half a year

CONTACTS AND LOCATIONS:
Overall Officials: yun liang, Principal Investigator — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No